CLINICAL TRIAL: NCT03938350
Title: Dialectical Behavior Therapy Skills Training for High-Risk African American Pregnant Women: Feasibility and Acceptability of Implementation in Prenatal Clinics
Brief Title: Dialectical Behavior Therapy for Pregnant Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Abigail Lott, Assistant Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00111022
Record Dates: First submitted 2019-05-02; First posted 2019-05-06 (Actual); Last update posted 2022-09-30 (Actual); Status verified 2022-09

CONDITIONS: Perinatal Depression
Keywords: Toxic stress; Maternal PTSD; Mindfulness-based intervention; Dialectical Behavior Therapy; Transgenerational transference of health disparities; Virtual intervention
MeSH Terms: interventions — Dialectical Behavior Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dialectical Behavior Therapy (DBT) Skills Training (Experimental): Participants in this group will receive 8 weeks of Dialectical Behavior Therapy (DBT) Skills Training.
  Interventions: Behavioral: Dialectical Behavior Therapy (DBT) Skills Training
- Treatment as Usual (No Intervention): Participants in this study arm will receive treatment as usual consisting of routine prenatal care with any mental health assessment, social work involvement or mental health service provision based on clinician referral or self-referral.

INTERVENTIONS:
Behavioral: Dialectical Behavior Therapy (DBT) Skills Training — Standard DBT skills training is a comprehensive intervention for emotion dysregulation that includes four skills modules: (1) mindfulness skills; (2) emotion regulation skills; (3) interpersonal effectiveness skills; and (4) distress tolerance skills designed to target adaptive skills deficits that define emotion dysregulation. The sessions will be delivered virtually via a HIPAA-compliant video platform.
  Arms: Dialectical Behavior Therapy (DBT) Skills Training

SUMMARY:
The cumulative effects of adverse childhood experiences (ACEs) can lead to prolonged activation of stress response systems, known as toxic stress. Toxic stress is increasingly recognized as an important contributor to socioeconomic and racial health disparities that emerge in early childhood and may persist across generations. African American women experience significant disparities in maternal and infant mortality, some of which may be attributable to toxic stress. The toxic stress response may increase risk factors for maternal and infant morbidity and mortality such as high-levels of stress hormones, high blood pressure, maternal PTSD and depression. Further, heightened maternal stress responses in pregnancy are associated with heightened infant stress responses, increasing the risk for the intergenerational transmission of toxic stress. Mindfulness-based interventions have demonstrated efficacy for a variety of mental health conditions, including depression and PTSD, are cost-effective, and scalable in diverse settings. Implementing mindfulness interventions for African American pregnant women with histories of ACEs and current depression and/or PTSD symptoms is novel and has the potential to interrupt the intergenerational cycle of toxic stress by improving maternal stress response and mental health. This study is a pilot, randomized controlled trial where participants will receive either Dialectical Behavior Therapy (DBT) Skills Training for 8 weeks (delivered virtually) or treatment as usual.

DETAILED DESCRIPTION:
The cumulative effects of adverse childhood experiences (ACEs), including trauma exposure, parent mental health problems, family dysfunction, and experiences of racism can lead to prolonged activation of stress response systems, known as toxic stress. Toxic stress can adversely influence maternal and childhood health. Increased numbers of ACEs are associated with negative birth outcomes such as decreased birth weight and gestational age at delivery. An intergenerational transmission of toxic stress has been evidenced in disruptions to children's hypothalamic pituitary adrenal (HPA)-axis functioning that result in life long health impacts. African American women are at increased risk for ACEs and similarly experience disparities in birth outcomes including low-birth weight and preterm birth. Many low-income, urban African American women are navigating the demands of pregnancy while confronting compounding chronic stressors, such as dangerous neighborhoods, lack of adequate and accessible public services, poverty, and the historical context of injustice, discrimination, and disadvantage. Although early life adversity can have serious consequences lasting across the lifespan and generations, interventions during critical periods such as pregnancy have the potential to prevent the intergenerational transmission of toxic stress and associated health disparities.

Prenatal mindfulness-based interventions have been shown to reduce depression, anxiety, and stress in pregnant women. Mindfulness is recommended as a culturally relevant intervention to reduce stress-related health disparities among African American and has been found to be feasible and acceptable to African American women. Further, mindfulness-based interventions are efficacious for a variety of mental health conditions and are cost-effective and scalable in diverse settings. Dialectical Behavior Therapy (DBT) Skills Training is a group format mindfulness-based intervention with demonstrated efficacy for increasing emotional regulation abilities and reducing depression and PTSD symptoms. DBT Skills Training has been adapted for trauma-exposed populations and is considered a transdiagnostic intervention for emotion dysregulation. Further, it is increasing being used with parents who have trauma histories and/or mental health problems. Adapting DBT skills for pregnant women with a history of ACEs and current depression and/or PTSD symptoms is novel and has the potential to interrupt the intergenerational cycle of toxic stress by improving maternal stress response, depression, and PTSD, thus reducing the risk of the intergenerational transmission of toxic stress.

This study will examine initial feasibility, acceptability, and effectiveness of an adapted 8-week DBT Skills Training group for mothers-to-be (DBTMTB) for low-income, African American pregnant women with a history of ACEs and current depression and PTSD symptoms to be delivered virtually. This adapted DBT Skills Training to the context of pregnancy will include specific pregnancy and parenting applications of DBT mindfulness and emotion regulation skills and opportunities to practice applying mindfulness and emotion regulation skills to enhance management of chronic stressors. The researchers posit that DBTMTB addresses important contributors to persistent birth outcome health disparities experienced by African American women and has the potential to reduce the cycle of toxic stress and transgenerational transference of disparities in health by improving pregnant women's mental health and stress response.

ELIGIBILITY:
Inclusion Criteria:

* Self-identify as African American/Black (includes African American/Black and another race)
* Able to read, speak, and understand English
* Adverse Childhood Experiences (ACE) score ≥ 4 from the Expanded ACE Questionnaire
* PHQ-9 score ≥ 9 or PC-PTSD-5 ≥ 3
* Within first or second trimester at time of recruitment
* Willing and able to participate in research assessments
* Willing and able to participate in a 8-week DBT Skills Training group for mothers-to-be (DBTMTB) Group
* Willing and able to provide informed consent

Exclusion Criteria:

* Presence of intellectual disability or actively displaying psychotic symptoms

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-10-16 (Actual); Primary Completion 2022-09-09 (Actual); Study Completion 2022-09-09 (Actual)

PRIMARY OUTCOMES:
Recruitment Rate | Baseline
  Feasibility of the intervention will be assessed by the number of women who agree to participate in the study, among those who are approached about participation.
Retention Rate | Week 8
  Feasibility of the intervention will be assessed by the number of participants completing the 8 week intervention.

SECONDARY OUTCOMES:
Acceptability of the Intervention | Week 8
  Acceptability of the intervention will be assessed through qualitative participant feedback. We will use a 25-item semi-structured interview to explore participants': (1) attitudes and beliefs related to the content of the intervention; (2) experiences with intervention components (e.g., facilitators' teaching skill, group interactions, and intervention exercises like role play/practices); and (3) barriers and facilitators for implementing the skills learned in the intervention in their daily life. Responses are in text form rather than on a pre-set scale.
Change in Patient Health Questionnaire (PHQ-9) Score | Baseline, Week 8
  The PHQ-9 is a 9-item self-report questionnaire developed to identify patients at risk for depression. Participants report how often they have been bothered by specific symptoms of depression on a scale of 0 (not at all) to 3 (nearly every day). Higher scores indicate greater symptoms of depression. A score of ≥ 9 indicates clinically significant symptoms.
Change in PTSD Checklist for Diagnostic and Statistical Manual of Mental Disorders (DSM)-5 (PCL-5) Score | Baseline, Week 8
  The PCL-5 instrument is a 20-item self-report measure that assesses DSM-5 symptoms of PTSD. Participants report how often they have been bothered by specific symptoms of PTSD on a scale of 0 (not at all) to 4 (extremely). The total symptom severity score ranges from 0 to 80. A provisional PTSD diagnosis can be made and a PCL-5 cut-point score of 33 is recommended.
Change in Difficulties in Emotion Regulation Scale (DERS) Score | Baseline, Week 8
  The DERS is a 36-item self-report measure that assesses 6 facets of emotion dysregulation. Participants report how much of the time they feel specific ways on a scale of 1 (almost never) to 5 (almost always). Totals scores range from 36 to 180 and higher scores indicate greater difficulties with emotion regulation.
Change in The Reflective Functioning Questionnaire (RFQ-8) Score | Baseline, Week 8
  The RFQ-8 is an 8-item self-report screener that assesses mentalizing or reflective functioning (understanding intentional mental states such as feelings, desires, and attitudes). Responses are given on a 7-point scale where 1 = strongly disagree and 7 = strongly agree (scoring is reversed for one item). Total raw scores range from 8 to 56 where higher scores indicate poorer reflective functioning.

CONTACTS AND LOCATIONS:
Overall Officials: Abigail Lott, PhD, Principal Investigator — Emory University; Briana Woods-Jaeger, PhD, Principal Investigator — Emory University
Locations (1):
- Grady Health System, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jones KA, Freijah I, Brennan SE, McKenzie JE, Bright TM, Fiolet R, Kamitsis I, Reid C, Davis E, Andrews S, Muzik M, Segal L, Herrman H, Chamberlain C. Interventions from pregnancy to two years after birth for parents experiencing complex post-traumatic stress disorder and/or with childhood experience of maltreatment. Cochrane Database Syst Rev. 2023 May 4;5(5):CD014874. doi: 10.1002/14651858.CD014874.pub2. PMID 37146219